CLINICAL TRIAL: NCT01393171
Title: Prospective Randomized Trial of Anterior Colporrhaphy Versus Cystocele Repair Using Polypropylene Mesh or Porcine Dermis
Brief Title: Anterior Colporrhaphy Versus Cystocele Repair Using Polypropylene Mesh or Porcine Dermis
Acronym: OARS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB4358; KPSC IRB 4358 (Other: Kaiser Permanente)
Record Dates: First submitted 2011-06-28; First posted 2011-07-13 (Estimated); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-10

CONDITIONS: Anterior Vaginal Wall Prolapse; Cystocele; Pelvic Organ Prolapse
Keywords: Anterior Vaginal Prolapse; Cystocele; Pelvic Organ Prolapse
MeSH Terms: conditions — Cystocele; Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Polypropylene Mesh (Active Comparator): Site-specific cystocele repair with polypropylene mesh augmentation
  Interventions: Device: Polypropylene mesh (Polyform by Boston Scientific)
- Anterior Colporrhaphy (Placebo Comparator): Anterior vaginal prolapse repair with anterior colporrhaphy with no graft.
  Interventions: Procedure: Anterior Colporrhaphy
- Porcine Dermis (Active Comparator): Site-specific cystocele repair with porcine dermis augmentation
  Interventions: Procedure: Porcine Dermis (Pelvicol by CRBard)

INTERVENTIONS:
Device: Polypropylene mesh (Polyform by Boston Scientific) — Site-specific cystocele repair with polypropylene mesh augmentation
  Other Names: Polyform by Boston Scientific
  Arms: Polypropylene Mesh
Procedure: Porcine Dermis (Pelvicol by CRBard) — Site-specific cystocele repair with porcine dermis augmentation
  Other Names: Pelvicol by CRBard
  Arms: Porcine Dermis
Procedure: Anterior Colporrhaphy — Anterior vaginal prolapse repair with suture.
  Other Names: Cystocele repair
  Arms: Anterior Colporrhaphy

SUMMARY:
The purpose of this study is to evaluate the success rate of cystocele repair using polypropylene mesh or porcine dermis compared to that of anterior colporrhaphy in a prospective randomized fashion. The study will be performed in a randomized, prospective, single-blinded fashion.

DETAILED DESCRIPTION:
Study participants will be recruited from the urogynecology clinic at Kaiser Permanente Medical Center Bellflower and San Diego. Clinical evaluation of each patient will include a standardized history, voiding diary, quality of life (UDI-6 & IIQ-7)10 and sexual function (PISQ-12)11-12 questionnaires (Attachment 1), urinalysis, gynecologic and pelvic organ prolapse quantification (POPQ) examinations. Patients will be randomized by a computer-generated randomization schedule, with allocation to either anterior colporrhaphy or site-specific cystocele repair with polypropylene mesh augmentation or site-specific cystocele repair with porcine dermis augmentation. The allocated treatment arm will be concealed in a sealed opaque envelope until the day of surgery. Patients will be given vaginal estrogen cream starting six weeks prior to surgery. Intravenous antibiotic prophylaxis will be given preoperatively and continued postoperatively for 24 hours. Vaginal infiltration will be performed with 0.25% bupivacaine and epinephrine (1:200,000) solution. Anterior colporrhaphy is performed by making a midline incision through the anterior vaginal mucosa, dissecting the vaginal epithelium from the underlying muscularis, and midline plication of the muscularis with No. 2-0 polydioxanone sutures (Ethicon, Somerville, NJ). The excess vaginal mucosa is then excised and the margins of the vagina reapproximated in the midline using No. 2-0 polyglactin (Vicryl) sutures. Patients who are randomized to polypropylene mesh or porcine dermis repair will undergo a site-specific defect repair of the vaginal muscularis with No. 2-0 polydioxanone sutures after midline vaginal incision and lateral dissection. A piece of the assigned material will be fashioned to fit the repaired space and anchored bilaterally to the arcus tendineus fascia pelvis with interrupted No. 2-0 polydioxanone sutures. Other operative procedures will be performed as indicated. TVT or TVT-O procedures (Gynecare Inc., Somerville, NJ) will be performed for stress urinary incontinence as previously described through a separate midurethral vaginal incision. The vagina will be packed for 24 hours. All patients will be discharged when they are able to ambulate and tolerate a solid diet and oral pain medication.

The two groups will be evaluated at 6 weeks, 6 months, 1 and 2 years after surgery. A trained clinical nurse/clinical fellow, whom has been proctored in performance of POP-Q exams, will perform postoperative POPQ staging in all patients. A research nurse blinded to the subject's group assignment will administer preoperative and postoperative quality of life and sexual function questionnaires. The primary outcome of this investigation will be postoperative anterior vaginal support. Anatomic success is defined as point Ba< -1. Secondary outcomes including hospital data, complications, subjective continence, quality of life and sexual function, and overall satisfaction with surgery, will also be compared.

ELIGIBILITY:
Inclusion Criteria:

* Stage 2 or > anterior vaginal prolapse requiring surgical correction.
* >18 years old
* willing to return for follow-up visits.

Exclusion Criteria:

* Less than stage II or > anterior vaginal prolapse,
* decline to participate,
* pregnant or contemplating future pregnancy,
* anti-incontinence procedure other than midurethral sling (ie, Burch colposuspension, pubovaginal sling, or needle suspension) is planned as part of their surgical procedures,
* any contra-indication to receiving mesh or porcine dermis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2018-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John N. Nguyen, MD, Principal Investigator — Kaiser Permanente
Locations (2):
- United States (2):
  - Kaiser Permanente, Downey, California
  - Kaiser Permanente, San Diego, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weber AM, Walters MD, Piedmonte MR, Ballard LA. Anterior colporrhaphy: a randomized trial of three surgical techniques. Am J Obstet Gynecol. 2001 Dec;185(6):1299-304; discussion 1304-6. doi: 10.1067/mob.2001.119081. PMID 11744900
- [Background] Altman D, Vayrynen T, Engh ME, Axelsen S, Falconer C; Nordic Transvaginal Mesh Group. Anterior colporrhaphy versus transvaginal mesh for pelvic-organ prolapse. N Engl J Med. 2011 May 12;364(19):1826-36. doi: 10.1056/NEJMoa1009521. PMID 21561348
- [Background] Simsiman AJ, Luber KM, Menefee SA. Vaginal paravaginal repair with porcine dermal reinforcement: correction of advanced anterior vaginal prolapse. Am J Obstet Gynecol. 2006 Dec;195(6):1832-6. doi: 10.1016/j.ajog.2006.07.005. Epub 2006 Sep 28. PMID 17010297
- [Result] Menefee SA, Dyer KY, Lukacz ES, Simsiman AJ, Luber KM, Nguyen JN. Colporrhaphy compared with mesh or graft-reinforced vaginal paravaginal repair for anterior vaginal wall prolapse: a randomized controlled trial. Obstet Gynecol. 2011 Dec;118(6):1337-1344. doi: 10.1097/AOG.0b013e318237edc4. PMID 22067717

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Polypropylene Mesh | Anterior Colporrhaphy | Porcine Dermis
Started (Oct 2005) | 36 | 32 | 31
Completed | 28 | 24 | 26
Not Completed | 8 | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Polypropylene Mesh | Anterior Colporrhaphy | Porcine Dermis | Total
Number analyzed (Participants) | 28 | 24 | 26 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (7) | 61 (11) | 60 (10) | 64 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 24 | 26 | 78
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Prospective Randomized Trial of Anterior Colporrhaphy Vs. Cystocele Repair Using Polypropylene Mesh or Porcine Dermis
Description: The primary outcome as the number of participants with optimal anterior vaginal support at two year defined as POPQ point Ba < -1.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Polypropylene Mesh | Anterior Colporrhaphy | Porcine Dermis
Number analyzed (Participants) | 28 | 24 | 26
Participants | 5 | 14 | 12

2. Secondary Outcome: Number of Participants With One or More Adverse Events at Two Years
Description: Number of participants with one or more adverse events at two years will also be compared between the three groups.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Polypropylene Mesh | Anterior Colporrhaphy | Porcine Dermis
Number analyzed (Participants) | 28 | 24 | 26
Participants | 7 | 4 | 5

3. Secondary Outcome: Number of Participants With Overall Failure
Description: Secondary Outcome Include:
  The number of participants with Overall Failure which includes subjective symptoms of vaginal bulge and POP-Q point of Ba > -1 on exam. This secondary outcome represents a composite outcome.
Time Frame: 2 year
Measure: Count of Participants; unit: Participants
Arm/Group | Polypropylene Mesh | Anterior Colporrhaphy | Porcine Dermis
Number analyzed (Participants) | 28 | 24 | 28
Participants | 1 | 3 | 3

4. Secondary Outcome: Change in Quality of Life Measured by the Pelvic Floor Distress Inventory 20 and Pelvic Floor Impact Questionnaire 7
Description: The difference in the Pelvic Floor Distress Inventory 20 (PFDI-20) and Pelvic Floor Impact Questionnaire 7 (PFIQ-7) score at 2 years compared to baseline values. The total score of each instrument ranges from 0 to 300 with higher scores indicating a greater degree of bother (ie, worse quality of life). The difference between baseline and 2-year scores were measured to account for differences in baseline scores among participants. A negative change in score indicates decreased bother after surgery and thus improved outcome; the greater the reduction in score, the greater reduction in bother and thus the better the outcome.
Time Frame: 2-year compared to baseline scores
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Polypropylene Mesh | Anterior Colporrhaphy | Porcine Dermis
Number analyzed (Participants) | 28 | 24 | 26
score on a scale
  PFDI-20 | -63 [-100 to 13] | -58 [-87 to -8] | -77 [-100 to 46]
  PFIQ-7 | -57 [-100 to -11] | -33 [-86 to -10] | -55 [-95 to 10]

5. Secondary Outcome: Change in Postoperative Sexual Function Measured by Pelvic Organ Prolapse/Urinary Incontinence Questionnaire 12
Description: The difference in Pelvic Organ Prolapse/Urinary Incontinence Questionnaire 12 (PISQ-12) scores at 24 months compared to baseline scores. The total score ranges from 0 to 48 with higher scores indicating better sexual function. The difference in PISQ-12 score was calculated to account for baseline variation in scores among participants. A positive change indicates improved sexual function while a negative change indicates worsened sexual function after surgery.
Time Frame: 2 year
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Polypropylene Mesh | Anterior Colporrhaphy | Porcine Dermis
Number analyzed (Participants) | 28 | 24 | 26
score on a scale | 0 [-28 to 36] | 0 [-32 to 16] | 1 [-35 to 24]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Polypropylene Mesh | Anterior Colporrhaphy | Porcine Dermis
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/24 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/24 | 0/26
Other Adverse Events (participants affected / at risk) | 7/28 | 4/24 | 5/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Polypropylene Mesh (N=28) | Anterior Colporrhaphy (N=24) | Porcine Dermis (N=26)
Vaginal implant exposure (Surgical and medical procedures) | 5 (5) | 0 (0) | 1 (1) — Number of patients with vaginal exposure of implant (mesh or porcine graft)
De novo stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2) — Number of participants with de novo stress urinary incontinence
De novo dyspareunia (Reproductive system and breast disorders) | 2 (2) | 3 (3) | 2 (2) — Number of participants with de novo dyspareunia

LIMITATIONS AND CAVEATS:
Small sample size that did not permit evaluation of differences between permanent mesh and xenografts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No